CLINICAL TRIAL: NCT00138151
Title: A Phase II Trial of Chemosensitization With Paclitaxel, 13-cis Retinoic Acid and Interferon Alpha-2b in Advanced Uterine Cervical Carcinoma
Brief Title: Isotretinoin, Interferon Alpha-2b, and Paclitaxel in Stage IV, Recurrent, or Persistent Cervical Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual and lack of study drug
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000433516; P30CA072720 (NIH); CINJ-100101 (Other: Cancer Institute of New Jersey); CINJ-3390 (Other: Cancer Institute of New Jersey); CINJ-NJ1703 (Other: Cancer Institute of New Jersey)
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-09

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; stage IVB cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Interferon alpha-2; Isotretinoin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel, 13-cis Retinoic Acid, and Interferon Alpha-2b (Experimental): * Cis-retinoic acid at a dose of 1 mg/kg/day PO qd days 1-4 of each cycle
  * Interferon alpha-2b at a dose of 6 mU/m2 SQ qd days 1-4 of each cycle
  * Paclitaxel 175 mg/m2 will be given on day 4. Cycles will be repeated every 21 days
  Interventions: Biological: recombinant interferon alpha-2b; Drug: isotretinoin; Drug: paclitaxel

INTERVENTIONS:
Biological: recombinant interferon alpha-2b — Interferon alpha-2b at a dose of 6 mU/m2 SQ qd days 1-4 of each cycle
Drug: isotretinoin — Cis-retinoic acid at a dose of 1 mg/kg/day PO qd days 1-4 of each cycle
Drug: paclitaxel — Paclitaxel 175 mg/m2 will be given on day 4. Cycles will be repeated every 21 days

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sometimes when chemotherapy is given, it does not stop the growth of tumor cells. The tumor is said to be resistant to chemotherapy. Giving isotretinoin and interferon alpha-2b together with paclitaxel may reduce drug resistance and allow the tumor cells to be killed.

PURPOSE: This phase II trial is studying how well giving isotretinoin and interferon alpha-2b together with paclitaxel works in treating patients with stage IV, recurrent, or persistent cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response in patients with stage IVB, recurrent, or persistent cervical cancer treated with isotretinoin, interferon alpha-2b, and paclitaxel.

OUTLINE: This is a multicenter study.

Patients receive oral isotretinoin and interferon alpha-2b subcutaneously once daily on days 1-4 and paclitaxel IV over 3 hours on day 4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 27-66 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and/or cytologically confirmed cervical cancer, meeting 1 of the following criteria:

  * Stage IVB disease
  * Recurrent disease
  * Persistent disease
* Patients previously treated with chemoradiotherapy as initial therapy must demonstrate disease progression
* Measurable disease by physical exam or radiographic studies
* Not amenable to chemoradiotherapy or surgery

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* WBC ≥ 3,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* SGOT and SGPT ≤ 2 times upper limit of normal
* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance ≥ 50 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity
* No active infection
* No medical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior interferon
* No other concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* At least 3 months since prior chemoradiotherapy (6 weeks for patients experiencing disease progression after completion of initial chemoradiotherapy)
* No other prior chemotherapy

Endocrine therapy

* No concurrent hormonal therapy for cancer

Radiotherapy

* See Disease Characteristics
* See Chemotherapy
* Recovered from prior radiotherapy
* No concurrent radiotherapy

Surgery

* Recovered from prior surgery
* No concurrent surgery for cancer

Other

* No prior retinoids
* No other concurrent anticancer therapy
* No other concurrent experimental agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2001-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Rodriguez, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (6):
- United States (6):
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - UMDNJ University Hospital, Newark, New Jersey
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 sites across New Jersey (2 academic medical centers and 2 community hospitals) from March 2001 through June 2009.
Period: Overall Study
Arm/Group | Paclitaxel, 13-cis Retinoic Acid, and Interferon Alpha-2b
Started | 33
Completed | 29
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel, 13-cis Retinoic Acid, and Interferon Alpha-2b
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 53.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete and Partial)
Description: All patients who receive at least 3 courses of protocol therapy will be considered evaluable for response of measurable disease.
Time Frame: 8 years
Population: Study was closed prematurely due to slow accrual and lack of study drug. Insufficient accrual to evaluate response rate.
Arm/Group | Paclitaxel, 13-cis Retinoic Acid, and Interferon Alpha-2b
Number analyzed (Participants) | 0

2. Secondary Outcome: The Effect of the Regimen on Bcl-2 Family Proteins in Biopsy Specimens and Correlation With Peripheral Blood Mononuclear Cell Bcl-2 Levels.
Time Frame: 8 years
Population: Study was closed prematurely due to slow accrual and lack of study drug. Insufficient accrual to evaluate response rate.
Arm/Group | Paclitaxel, 13-cis Retinoic Acid, and Interferon Alpha-2b
Number analyzed (Participants) | 0

3. Secondary Outcome: The Effect of the Regimen on Raf-1 Kinase Phosphorylation in Biopsy Specimens.
Time Frame: 8 years
Population: Study was closed prematurely due to slow accrual and lack of study drug. Insufficient accrual to evaluate response rate.
Arm/Group | Paclitaxel, 13-cis Retinoic Acid, and Interferon Alpha-2b
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 8 years
Arm/Group | Paclitaxel, 13-cis Retinoic Acid, and Interferon Alpha-2b
Serious Adverse Events (participants affected / at risk) | 18/33
Other Adverse Events (participants affected / at risk) | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel, 13-cis Retinoic Acid, and Interferon Alpha-2b (N=33)
Hyponatremia (Investigations) | 2 (2)
Abdominal pain (General disorders) | 3 (3)
Infection without neutropenia (Infections and infestations) | 8 (9)
Fatigue (General disorders) | 1 (1)
Thrombosis/embolism (Blood and lymphatic system disorders) | 2 (2)
Fever in the absence of neutropenia where neutropenia is defined as AGC <1.0 x 10e9/L (General disorders) | 4 (4)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fistula or GU fistula (e.g., vaginal, vesicovaginal) (Renal and urinary disorders) | 1 (1)
Ureteral obstruction (Renal and urinary disorders) | 1 (1)
Edema (Vascular disorders) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 3 (6)
Dehydration (Gastrointestinal disorders) | 2 (2)
Depressed level of consciousness - somnolence (Nervous system disorders) | 1 (1)
Vaginal bleeding (Blood and lymphatic system disorders) | 1 (1)
Hyperkalemia (Investigations) | 1 (1)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (other) - back pain (General disorders) | 4 (5)
Congestive heart failure (Cardiac disorders) | 1 (2)
Dypsnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection/Febrile Neutropenia (Infections and infestations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary other - respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypocalcemia (Investigations) | 1 (1)
Mood alteration - anxiety, agitation (Psychiatric disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hematuria (in the absence of vaginal bleeding) (Blood and lymphatic system disorders) | 1 (1)
Elevated ammonia level (Investigations) | 1 (1)
Death (General disorders) | 1 (1)
Hypokalemia (Investigations) | 2 (2)
Hypomagnesemia (Investigations) | 1 (1)
Fracture - neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical spinal cord compression (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Change in mental status (Nervous system disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Rectal bleeding/hematochezia (Blood and lymphatic system disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel, 13-cis Retinoic Acid, and Interferon Alpha-2b (N=33)
Nausea (Gastrointestinal disorders) | 16 (33)
Vomiting (Gastrointestinal disorders) | 12 (15)
Diarrhea, patients without colostomy (Gastrointestinal disorders) | 11 (15)
Constipation (Gastrointestinal disorders) | 10 (13)
Anorexia (Gastrointestinal disorders) | 7 (9)
Gastrointestinal - other (Gastrointestinal disorders) | 6 (6)
Dehydration (Gastrointestinal disorders) | 3 (3)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 2 (2)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies, if specified in the protocol (Gastrointestinal disorders) | 2 (2)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 19 (31)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 16 (24)
Rigors, chills (General disorders) | 8 (13)
Constitutional Symptoms-Other (Specify,_____) (General disorders) | 4 (6)
Pain-Other (Specify,___) (General disorders) | 17 (31)
Headache (General disorders) | 7 (8)
Abdominal pain or cramping (Gastrointestinal disorders) | 6 (6)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 6 (9)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (22)
Dermatology/Skin-Other (Specify,_____) (Skin and subcutaneous tissue disorders) | 3 (6)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 9 (16)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 9 (33)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 7 (28)
Blood/Bone Marrow-Other (Specify,_____) (Blood and lymphatic system disorders) | 3 (4)
Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol (Blood and lymphatic system disorders) | 2 (2)
Neuropathy-sensory (Nervous system disorders) | 10 (17)
Mood alteration-anxiety, agitation (Psychiatric disorders) | 4 (4)
Mood alteration-depression (Psychiatric disorders) | 4 (4)
Dizziness/lightheadedness (Nervous system disorders) | 3 (3)
Insomnia (Nervous system disorders) | 3 (3)
Neurology-Other (Specify,______) (Nervous system disorders) | 2 (2)
Renal/Genitourinary-Other (Specify,____) (Renal and urinary disorders) | 4 (4)
Urinary frequency/urgency (Renal and urinary disorders) | 4 (5)
Dysuria (painful urination) (Renal and urinary disorders) | 2 (2)
Ureteral obstruction (Renal and urinary disorders) | 2 (2)
Hypertriglyceridemia (Investigations) | 3 (3)
Hypercholesterolemia (Investigations) | 2 (2)
Hyperglycemia (Investigations) | 2 (2)
Hyperuricemia (Investigations) | 2 (2)
Hypokalemia (Investigations) | 2 (2)
Edema (Vascular disorders) | 6 (7)
Hypertension (Cardiac disorders) | 2 (2)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal-Other (Specify,______) (Musculoskeletal and connective tissue disorders) | 3 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 2 (2)
Infection without neutropenia (Infections and infestations) | 2 (3)
Infection/Febrile Neutropenia-Other (Specify,____) (Infections and infestations) | 2 (3)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2)
Hot flashes/flushes (Endocrine disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes